CLINICAL TRIAL: NCT06707233
Title: Y-90 Selective Internal Radiation Therapy for Unresectable Hepatocellular Carcinoma Larger Than 7cm: a Prospective, Single Arm Trial
Brief Title: Y-90 SIRT for Unresectable HCC Larger Than 7cm
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-17
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma Non-Resectable
Keywords: Hepatocellular Carcinoma; yttrium-90; selective internal radiation therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sirtuins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SIRT (Experimental): Patients will receive SIRT treatment
  Interventions: Procedure: SIRT

INTERVENTIONS:
Procedure: SIRT — The patients will receive 1-2 sessions of SIRT.

SUMMARY:
This is a phase II clinical study to evaluate the efficacy and safety of SIRT in patients with HCC greater than 7 cm. After enrollment, patients received yttrium-90 selective internal radiation therapy. The primary endpoint of the study is objective reponse rate (ORR) as assessed by mRECIST. Secondary endpoints were: objective response rate (ORR) as assessed by RECIST 1.1, disease control rate (DCR), progression-free survival (PFS), time to response (TTR), duration of response (DOR), overall survival (OS), and safety (incidence and severity of adverse events).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed or clinically diagnosed HCC
* Unresectable HCC as assessed by a team of surgeons
* The largest tumor size > 7 cm
* Tumor recurrence after curative treatment (hepatectomy or ablation) is eligible for enrollment
* At least one measurable intrahepatic target lesion
* Appropriate for SIRT treatment after evaluation (including SPECT/CT evaluation after arterial perfusion with 99Tc-MAA)
* Child-Pugh score ≤ 7
* ECOG PS ≤ 1
* Adequate organ and hematologic function with platelet count ≥75×10^9/L, leukocyte >3.0×10^9/L, Neutrophil count ≥1.5×10^9/L, haemoglobin ≥85 g/L, ALT and AST≤5×ULN, creatinine≤1.5×ULN, and prolongation of prothrombin time ≤4 seconds
* life expectancy of at least 6 months

Exclusion Criteria:

* Macrovascular invasion or extrahepatic metastasis
* Decompensated liver function, including: ascites, bleeding from gastroesophageal varices, and hepatic encephalopathy
* Organ (heart and kidneys) dysfunction
* History of other malignancies
* Uncontrollable infection
* History of organ or cells transplantation
* History of HIV
* Pregnant or lactating patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) per mRECIST | 3 years
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to mRECIST

SECONDARY OUTCOMES:
Objective response rate (ORR) per RECIST 1.1 | 3 years
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to RECIST 1.1
Disease control rate (DCR) | 3 years
  The proportion of patients with the best response of CR, PR, or stable disease (SD) according to mRECIST and RECIST 1.1
Progression free survival (PFS) | 3 years
  The time from date of treatment initiation until the first occurrence of disease progression (according to mRECIST and RECIST 1.1) or death due to any cause, whichever occurs first.
time to response (TTR) | 3 years
  The time from treatment initiation to first tumour remission (mRECIST and RECIST 1.1)
Duration of response (DOR) | 3 years
  Time from first tumor response to first disease progression (mRECIST and RECIST 1.1 assessment) or death from any cause (whichever occurs first)
Overall survival (OS) | 4 years
  The time from date of treatment initiation to death due to any cause
Adverse Events (AEs) | 3 years
  Number of patients with AEs assessed by Common Terminology Criteria for Adverse Events v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided